CLINICAL TRIAL: NCT06614231
Title: Prospective Phase II Trial of Neoajuvant Tislelizumab Combined with Chemotherapy for Initially Unresectable Stage IIIA/N2 Non-small Cell Lung Cancer
Brief Title: Neoajuvant Tislelizumab Combined with Chemotherapy for Initially Unresectable Stage IIIA/N2 Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Hou, Professor of Medicine, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-446-01
Record Dates: First submitted 2024-09-12; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: NSCLC, Stage IIIA; NSCLC (non-small Cell Lung Cancer)
Keywords: Unresectable stage III NSCLC; Tirellizumab; Neoadjuvant treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab (Experimental): Tislelizumab 200mg Q3W
  Interventions: Drug: Tislelizumab Combined With Chemotherapy

INTERVENTIONS:
Drug: Tislelizumab Combined With Chemotherapy — Tislelizumab 200mg Q3W，Platinum-containing dual drug chemotherapy
  Other Names: Platinum-containing

SUMMARY:
To investigate the efficacy and safety of neoadjuvant treatment with Tislelizumab combined with chemotherapy for initially unresectable N2/III non-small cell lung cancer.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, single-center phase II clinical trial to investigate the efficacy and safety of neoadjuvant treatment with tirilizumab in combination with chemotherapy in patients with initially inoperable stage III/N2 non-small cell lung cancer.

Patients with stage III/N2 non-small cell lung cancer that is initially inoperable and clearly staged and meets the enrollment criteria will receive 3 cycles of tirilizumab (200 mg) in combination with chemotherapy and will be evaluated by imaging of their tumor status. After MDT evaluation patients will either undergo surgery or be withdrawn from the study and receive a combination of radiotherapy and chemotherapy, with postoperative adjuvant therapy at the discretion of the physician. The primary endpoint of this study is the surgical conversion rate; secondary endpoints include MPR, pCR, safety, and EFS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with initially untreated, unresectable stage III NSCLC (according to the International Association for the Study of Lung Cancer IASLC 8th Thoracic Tumor Stage) with non-small cell lung cancer
2. All patients received baseline PET/CT (or neck, upper thoracic and abdominal CT+ cranial MR) for clinical staging
3. Cytology/histology (mediastinoscopy or EBUS, etc.) confirmed N2 non-small cell lung cancer
4. For non-squamous cell carcinoma patients, if EGFR/ALK mutation status is unknown, tissue samples should be provided for EGFR/ALK gene testing before enrollment; For patients with squamous cell carcinoma, if EGFR/ALK mutation status is unknown, testing is not required during screening
5. ECOG (Performance status, PS) score 0-1
6. Hematology testings meet the following requirements

   * neutrophil ≥1.5*109/L
   * Platelets ≥100*109/L
   * Hemoglobin > 9.0 g/dL
   * Serum creatinine ≤1.5ULN or creatinine clearance (Ccr) ≥40mL/min
   * AST/ALT≤ 3ULN
   * Total bilirubin ≤1.5ULN
   * FEV1≥1.2L or > 40% of the estimated value
   * INR/APTT within normal range
7. The patient is over 18 years old
8. Measurable lesions (according to the RECIST 1.1 version)
9. Subject must understand and voluntarily sign informed consent prior to any study-related evaluation

Exclusion Criteria

1. The patient presents with a confirmed or suspected autoimmune disorder.

   * Note: Patients with vitiligo, type I diabetes mellitus, or Hashimoto's thyroiditis who are hypothyroid but require only hormone replacement therapy may be included in the study if there are no obvious signs of relapse
2. Patients must have undergone systemic corticosteroid treatment (≥10mg prednisolone [or equivalent]/day) or received other immunosuppressive medications within 14 days prior to enrollment.

   * Note: Inhaled or topical corticosteroids and adrenal hormone replacement therapy (≥10mg prednisolone [or equivalent]/day) can also be accepted for individuals lacking clear evidence of autoimmune disorders
3. Patients with grade 3 or 4 interstitial lung disease
4. Have other malignant tumors and need anti-tumor therapy
5. Patients with previous malignancies (except skin malignancies other than melanoma, and in situ cancers of the following sites (bladder, stomach, colorectal, endometrial, cervix, melanoma, or breast) were not included in the study. Unless the malignancy has been in complete remission for two years or more and no additional antitumor therapy is required during the study period
6. The investigator believes that the patient is medically, psychologically, or physically incapable of completing this study or of understanding the patient handbook information
7. Previously received anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA, and other drugs targeting T-cell co-stimulation or immune regulatory pathways
8. Presence of active Hepatitis B or C
9. HIV-positive or diagnosed with Acquired Immune Deficiency Disease (AIDS)
10. Allergy to the study drug
11. Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2028-09-08 (Estimated); Study Completion 2028-09-08 (Estimated)

PRIMARY OUTCOMES:
Surgical conversion rate | Within 4-6 weeks (+7 days) after the third cycle of Tislelizumab combined with chemotherapy
  After 3 cycles of Tislelizumab combined with chemotherapy, the number of patients who underwent surgical resection/number of patients enrolled

SECONDARY OUTCOMES:
Major pathologic response(MPR) | Within one week after surgery
  Less than 10% of tumor cells remained in the pathological excision specimen
Pathologic Complete response（pCR） | Within one week after surgery
  No tumor cells were observed in pathological excision specimens

IPD SHARING:
Plan to Share IPD: Yes
publish an article